CLINICAL TRIAL: NCT04347811
Title: Systematic Trial Of PrevenTing Healthcare Employee Burnout: Using Reflection & Nourishment
Brief Title: Use of Death Cafes to Prevent Burnout in ICU Healthcare Employees
Acronym: STOPTHEBURN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: Spirit of Charity Foundation - University Medical Center (Unknown)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-908
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Burnout; Burnout, Professional; Burnout, Psychological; Anxiety; Depression
Keywords: Critical Care; Nurses; Physicians; Healthcare Workers; Death; Grief; Stress, Psychological; Occupational Stress; Behavioral Symptoms; Coping Skills; Clinical Trial
MeSH Terms: conditions — Burnout, Psychological; Burnout, Professional; Anxiety Disorders; Depression; Death; Stress, Psychological; Occupational Stress; Behavioral Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Death Cafe Arm (Experimental): Participants undergo biweekly Death Café sessions hosted by a trained psychotherapist for 3 months.
  Interventions: Behavioral: Death Cafe
- Control Arm (No Intervention): Participants do not undergo biweekly Death Café sessions hosted by a trained psychotherapist for 3 months.

INTERVENTIONS:
Behavioral: Death Cafe — Death Cafés are a specific form of debriefing that focuses on discussing death, dying, loss, and illness. Nourishment in the form of cake is provided. These sessions may allow for reflection on distressing patient events while developing a sense of community and collaboration among hospital employees.
  Arms: Death Cafe Arm

SUMMARY:
Burnout affects a significant number of healthcare employees and leads to worsened mental health, increased job turnover, and patient safety events. Those caring for critically ill patients may be especially susceptible due to high patient mortality, long hours, and regular encounters with traumatic and ethical issues. Preliminary studies suggest that debriefing opportunities may reduce burnout through reflection on distressing patient events, enhancement of social support, and interprofessional collaboration. Death Cafés are a specific form of debriefing that focus on discussing death, dying, loss, and illness.

The purpose of this study is to evaluate whether biweekly Death Cafe group debriefing sessions can prevent burnout in ICU physicians and staff.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, nurses, pharmacists, or therapists working in the Intensive Care Unit and have worked for the full-time equivalent of at least 1 week in the preceding 4 weeks

Exclusion Criteria:

* Not physicians, nurses, pharmacists, or therapists
* Have worked less than the full-time equivalent of at least 1 week in the preceding 4 weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Differences in Burnout as measured by the Maslach Burnout Inventory Score (MBI). | At the time of enrollment and at 1 month, 3 months, 6 months after enrollment
  This is a validated 22-item, self-reported questionnaire that asks respondents to indicate on a 7 point Likert scale the frequency of certain feelings related to their job. Presence of burnout is defined by high values of depersonalization and emotional exhaustion with low values for personal accomplishment. Changes in mean scores between groups and within groups over time will be assessed.

SECONDARY OUTCOMES:
Differences in Depression as measured by the Patient Health Questionnaire 8 (PHQ-8) | At the time of enrollment and at 1 month, 3 months, 6 months after enrollment
  This is an 8 question validated questionnaire that asks respondents to indicate the frequency with which they have experienced certain symptoms consistent with depression. Higher scores mean higher frequency of depression symptoms, and a score of 10 or higher will be considered to indicate clinically significant depression. Changes in mean scores between groups and within groups over time will be assessed.
Differences in Anxiety as measured by the Generalized Anxiety Disorder 7 Scale (GAD-7) | At the time of enrollment and at 1 month, 3 months, 6 months after enrollment
  This is a 7 question validated questionnaire that asks respondents to indicate the frequency with which they have experienced certain symptoms consistent with anxiety. Higher scores mean higher frequency of anxiety symptoms, and a score of 10 or higher will be considered to indicate clinically significant anxiety. Changes in mean scores between groups and within groups over time will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie E Bateman, MD, Principal Investigator — Tulane University School of Medicine; Joshua Denson, MD, Principal Investigator — Tulane University School of Medicine
Locations (4):
- United States (4):
  - Tulane Medical Center, New Orleans, Louisiana
  - University Medical Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maslach C, Schaufeli WB, Leiter MP. Job burnout. Annu Rev Psychol. 2001;52:397-422. doi: 10.1146/annurev.psych.52.1.397. PMID 11148311
- [Background] Hammer R, Ravindran N, Nielsen N. Can Death Cafes resuscitate morale in hospitals? Med Humanit. 2021 Mar;47(1):2-3. doi: 10.1136/medhum-2018-011607. Epub 2019 Jan 19. PMID 30661041
- [Background] Rodrigues H, Cobucci R, Oliveira A, Cabral JV, Medeiros L, Gurgel K, Souza T, Goncalves AK. Burnout syndrome among medical residents: A systematic review and meta-analysis. PLoS One. 2018 Nov 12;13(11):e0206840. doi: 10.1371/journal.pone.0206840. eCollection 2018. PMID 30418984
- [Background] Elmariah H, Thomas S, Boggan JC, Zaas A, Bae J. The Burden of Burnout. Am J Med Qual. 2017 Mar/Apr;32(2):156-162. doi: 10.1177/1062860615625802. Epub 2016 Jul 9. PMID 26917807
- [Background] Holmes EG, Connolly A, Putnam KT, Penaskovic KM, Denniston CR, Clark LH, Rubinow DR, Meltzer-Brody S. Taking Care of Our Own: A Multispecialty Study of Resident and Program Director Perspectives on Contributors to Burnout and Potential Interventions. Acad Psychiatry. 2017 Apr;41(2):159-166. doi: 10.1007/s40596-016-0590-3. Epub 2016 Jul 19. PMID 27436125
- [Background] Thrush CR, Guise JB, Gathright MM, Messias E, Flynn V, Belknap T, Thapa PB, Williams DK, Nada EM, Clardy JA. A One-Year Institutional View of Resident Physician Burnout. Acad Psychiatry. 2019 Aug;43(4):361-368. doi: 10.1007/s40596-019-01043-9. Epub 2019 Feb 28. PMID 30820845
- [Background] Thomas NK. Resident burnout. JAMA. 2004 Dec 15;292(23):2880-9. doi: 10.1001/jama.292.23.2880. PMID 15598920
- [Background] Ishak WW, Lederer S, Mandili C, Nikravesh R, Seligman L, Vasa M, Ogunyemi D, Bernstein CA. Burnout during residency training: a literature review. J Grad Med Educ. 2009 Dec;1(2):236-42. doi: 10.4300/JGME-D-09-00054.1. PMID 21975985
- [Background] Dzau VJ, Kirch DG, Nasca TJ. To Care Is Human - Collectively Confronting the Clinician-Burnout Crisis. N Engl J Med. 2018 Jan 25;378(4):312-314. doi: 10.1056/NEJMp1715127. No abstract available. PMID 29365296
- [Background] Moss M, Good VS, Gozal D, Kleinpell R, Sessler CN. An Official Critical Care Societies Collaborative Statement-Burnout Syndrome in Critical Care Health-care Professionals: A Call for Action. Chest. 2016 Jul;150(1):17-26. doi: 10.1016/j.chest.2016.02.649. PMID 27396776
- [Background] Filho FA, Rodrigues MCS, Cimiotti JP. Burnout in Brazilian Intensive Care Units: A Comparison of Nurses and Nurse Technicians. AACN Adv Crit Care. 2019 Spring;30(1):16-21. doi: 10.4037/aacnacc2019222. PMID 30842069
- [Background] Zhang XC, Huang DS, Guan P; SUBLIN Study Team. Job burnout among critical care nurses from 14 adult intensive care units in Northeastern China: a cross-sectional survey. BMJ Open. 2014 Jun 19;4(6):e004813. doi: 10.1136/bmjopen-2014-004813. PMID 24948747
- [Background] Guntupalli KK, Wachtel S, Mallampalli A, Surani S. Burnout in the intensive care unit professionals. Indian J Crit Care Med. 2014 Mar;18(3):139-43. doi: 10.4103/0972-5229.128703. PMID 24701063
- [Background] Ahmadi O, Azizkhani R, Basravi M. Correlation between workplace and occupational burnout syndrome in nurses. Adv Biomed Res. 2014 Jan 24;3:44. doi: 10.4103/2277-9175.125751. eCollection 2014. PMID 24627852
- [Background] Poncet MC, Toullic P, Papazian L, Kentish-Barnes N, Timsit JF, Pochard F, Chevret S, Schlemmer B, Azoulay E. Burnout syndrome in critical care nursing staff. Am J Respir Crit Care Med. 2007 Apr 1;175(7):698-704. doi: 10.1164/rccm.200606-806OC. Epub 2006 Nov 16. PMID 17110646
- [Background] Embriaco N, Papazian L, Kentish-Barnes N, Pochard F, Azoulay E. Burnout syndrome among critical care healthcare workers. Curr Opin Crit Care. 2007 Oct;13(5):482-8. doi: 10.1097/MCC.0b013e3282efd28a. PMID 17762223
- [Background] Johnson-Coyle L, Opgenorth D, Bellows M, Dhaliwal J, Richardson-Carr S, Bagshaw SM. Moral distress and burnout among cardiovascular surgery intensive care unit healthcare professionals: A prospective cross-sectional survey. Can J Crit Care Nurs. 2016 Jan;27(4):27-36. PMID 29786979
- [Background] Edmondson EK, Kumar AA, Smith SM. Creating a Culture of Wellness in Residency. Acad Med. 2018 Jul;93(7):966-968. doi: 10.1097/ACM.0000000000002250. PMID 29668521
- [Background] Lu DW, Dresden S, McCloskey C, Branzetti J, Gisondi MA. Impact of Burnout on Self-Reported Patient Care Among Emergency Physicians. West J Emerg Med. 2015 Dec;16(7):996-1001. doi: 10.5811/westjem.2015.9.27945. Epub 2015 Dec 11. PMID 26759643
- [Background] Schwarzkopf D, Ruddel H, Thomas-Ruddel DO, Felfe J, Poidinger B, Matthaus-Kramer CT, Hartog CS, Bloos F. Perceived Nonbeneficial Treatment of Patients, Burnout, and Intention to Leave the Job Among ICU Nurses and Junior and Senior Physicians. Crit Care Med. 2017 Mar;45(3):e265-e273. doi: 10.1097/CCM.0000000000002081. PMID 27776092
- [Background] Sklar DP. Fostering Student, Resident, and Faculty Wellness to Produce Healthy Doctors and a Healthy Population. Acad Med. 2016 Sep;91(9):1185-8. doi: 10.1097/ACM.0000000000001298. No abstract available. PMID 27576028
- [Background] Shanafelt TD, Balch CM, Bechamps G, Russell T, Dyrbye L, Satele D, Collicott P, Novotny PJ, Sloan J, Freischlag J. Burnout and medical errors among American surgeons. Ann Surg. 2010 Jun;251(6):995-1000. doi: 10.1097/SLA.0b013e3181bfdab3. PMID 19934755
- [Background] Dewa CS, Loong D, Bonato S, Trojanowski L, Rea M. The relationship between resident burnout and safety-related and acceptability-related quality of healthcare: a systematic literature review. BMC Med Educ. 2017 Nov 9;17(1):195. doi: 10.1186/s12909-017-1040-y. PMID 29121895
- [Background] Baer TE, Feraco AM, Tuysuzoglu Sagalowsky S, Williams D, Litman HJ, Vinci RJ. Pediatric Resident Burnout and Attitudes Toward Patients. Pediatrics. 2017 Mar;139(3):e20162163. doi: 10.1542/peds.2016-2163. PMID 28232639
- [Background] Block L, Wu AW, Feldman L, Yeh HC, Desai SV. Residency schedule, burnout and patient care among first-year residents. Postgrad Med J. 2013 Sep;89(1055):495-500. doi: 10.1136/postgradmedj-2012-131743. Epub 2013 Jul 14. PMID 23852828
- [Background] Kang EK, Lihm HS, Kong EH. Association of intern and resident burnout with self-reported medical errors. Korean J Fam Med. 2013 Jan;34(1):36-42. doi: 10.4082/kjfm.2013.34.1.36. Epub 2013 Jan 28. PMID 23372904
- [Background] Kiymaz D, Koc Z. Identification of factors which affect the tendency towards and attitudes of emergency unit nurses to make medical errors. J Clin Nurs. 2018 Mar;27(5-6):1160-1169. doi: 10.1111/jocn.14148. Epub 2018 Feb 21. PMID 29076206
- [Background] Mohammadi M, Peyrovi H, Mahmoodi M. The Relationship Between Professional Quality of Life and Caring Ability in Critical Care Nurses. Dimens Crit Care Nurs. 2017 Sep/Oct;36(5):273-277. doi: 10.1097/DCC.0000000000000263. PMID 28777112
- [Background] Passalacqua SA, Segrin C. The effect of resident physician stress, burnout, and empathy on patient-centered communication during the long-call shift. Health Commun. 2012;27(5):449-56. doi: 10.1080/10410236.2011.606527. Epub 2011 Oct 4. PMID 21970629
- [Background] Prins JT, van der Heijden FM, Hoekstra-Weebers JE, Bakker AB, van de Wiel HB, Jacobs B, Gazendam-Donofrio SM. Burnout, engagement and resident physicians' self-reported errors. Psychol Health Med. 2009 Dec;14(6):654-66. doi: 10.1080/13548500903311554. PMID 20183538
- [Background] West CP, Tan AD, Habermann TM, Sloan JA, Shanafelt TD. Association of resident fatigue and distress with perceived medical errors. JAMA. 2009 Sep 23;302(12):1294-300. doi: 10.1001/jama.2009.1389. PMID 19773564
- [Background] Fahrenkopf AM, Sectish TC, Barger LK, Sharek PJ, Lewin D, Chiang VW, Edwards S, Wiedermann BL, Landrigan CP. Rates of medication errors among depressed and burnt out residents: prospective cohort study. BMJ. 2008 Mar 1;336(7642):488-91. doi: 10.1136/bmj.39469.763218.BE. Epub 2008 Feb 7. PMID 18258931
- [Background] West CP, Huschka MM, Novotny PJ, Sloan JA, Kolars JC, Habermann TM, Shanafelt TD. Association of perceived medical errors with resident distress and empathy: a prospective longitudinal study. JAMA. 2006 Sep 6;296(9):1071-8. doi: 10.1001/jama.296.9.1071. PMID 16954486
- [Background] Shanafelt TD, Bradley KA, Wipf JE, Back AL. Burnout and self-reported patient care in an internal medicine residency program. Ann Intern Med. 2002 Mar 5;136(5):358-67. doi: 10.7326/0003-4819-136-5-200203050-00008. PMID 11874308
- [Background] Walsh AL, Lehmann S, Zabinski J, Truskey M, Purvis T, Gould NF, Stagno S, Chisolm MS. Interventions to Prevent and Reduce Burnout Among Undergraduate and Graduate Medical Education Trainees: a Systematic Review. Acad Psychiatry. 2019 Aug;43(4):386-395. doi: 10.1007/s40596-019-01023-z. Epub 2019 Feb 1. PMID 30710229
- [Background] Jarden RJ, Sandham M, Siegert RJ, Koziol-McLain J. Strengthening workplace well-being: perceptions of intensive care nurses. Nurs Crit Care. 2019 Jan;24(1):15-23. doi: 10.1111/nicc.12386. Epub 2018 Sep 21. PMID 30240098
- [Background] Govindan M, Keefer P, Sturza J, Stephens MR, Malas N. Empowering Residents to Process Distressing Events: A Debriefing Workshop. MedEdPORTAL. 2019 Feb 27;15:10809. doi: 10.15766/mep_2374-8265.10809. PMID 30931388
- [Background] McDermott A, Brook I, Ben-Isaac E. Peer-Debriefing After Distressing Patient Care Events: A Workshop for Pediatric Residents. MedEdPORTAL. 2017 Sep 5;13:10624. doi: 10.15766/mep_2374-8265.10624. PMID 30800825
- [Background] Hellyar M, Madani C, Yeaman S, O'Connor K, Kerr KM, Davidson JE. Case Study Investigation Decreases Burnout While Improving Interprofessional Teamwork, Nurse Satisfaction, and Patient Safety. Crit Care Nurs Q. 2019 Jan/Mar;42(1):96-105. doi: 10.1097/CNQ.0000000000000243. PMID 30507670
- [Background] Lederer W, Kinzl JF, Traweger C, Dosch J, Sumann G. Fully developed burnout and burnout risk in intensive care personnel at a university hospital. Anaesth Intensive Care. 2008 Mar;36(2):208-13. doi: 10.1177/0310057X0803600211. PMID 18361012
- [Background] Ricou B, Gigon F, Durand-Steiner E, Liesenberg M, Chemin-Renais C, Merlani P, Delaloye S. Initiative for Burnout of ICU Caregivers: Feasibility and Preliminary Results of a Psychological Support. J Intensive Care Med. 2020 Jun;35(6):562-569. doi: 10.1177/0885066618768223. Epub 2018 Apr 11. PMID 29642743
- [Background] Browning ED, Cruz JS. Reflective Debriefing: A Social Work Intervention Addressing Moral Distress among ICU Nurses. J Soc Work End Life Palliat Care. 2018 Jan-Mar;14(1):44-72. doi: 10.1080/15524256.2018.1437588. Epub 2018 Feb 28. PMID 29488856
- [Background] Eagle S, Creel A, Alexandrov A. The effect of facilitated peer support sessions on burnout and grief management among health care providers in pediatric intensive care units: a pilot study. J Palliat Med. 2012 Nov;15(11):1178-80. doi: 10.1089/jpm.2012.0231. Epub 2012 Aug 21. PMID 22909377
- [Background] Colville GA, Smith JG, Brierley J, Citron K, Nguru NM, Shaunak PD, Tam O, Perkins-Porras L. Coping With Staff Burnout and Work-Related Posttraumatic Stress in Intensive Care. Pediatr Crit Care Med. 2017 Jul;18(7):e267-e273. doi: 10.1097/PCC.0000000000001179. PMID 28459762
- [Background] Schmidt M, Haglund K. Debrief in Emergency Departments to Improve Compassion Fatigue and Promote Resiliency. J Trauma Nurs. 2017 Sep/Oct;24(5):317-322. doi: 10.1097/JTN.0000000000000315. PMID 28885522
- [Background] Leff V, Klement A, Galanos A. A Successful Debrief Program for House Staff. J Soc Work End Life Palliat Care. 2017 Apr-Sep;13(2-3):87-90. doi: 10.1080/15524256.2017.1314234. Epub 2017 Apr 20. PMID 28426397
- [Background] Klein SD, Bucher HU, Hendriks MJ, Baumann-Holzle R, Streuli JC, Berger TM, Fauchere JC, On Behalf Of The Swiss Neonatal End-Of-Life Study Group. Sources of distress for physicians and nurses working in Swiss neonatal intensive care units. Swiss Med Wkly. 2017 Aug 3;147:w14477. doi: 10.4414/smw.2017.14477. eCollection 2017. PMID 28804867
- [Background] Ziegelstein RC. Creating Structured Opportunities for Social Engagement to Promote Well-Being and Avoid Burnout in Medical Students and Residents. Acad Med. 2018 Apr;93(4):537-539. doi: 10.1097/ACM.0000000000002117. PMID 29280756
- [Background] Abrams MP. Improving Resident Well-Being and Burnout: The Role of Peer Support. J Grad Med Educ. 2017 Apr;9(2):264. doi: 10.4300/JGME-D-16-00805.1. No abstract available. PMID 28439373
- [Background] Miles L, Corr CA. Death Cafe. Omega (Westport). 2017 Jun;75(2):151-165. doi: 10.1177/0030222815612602. Epub 2015 Oct 29. PMID 28490282
- [Background] Nelson KE, Wright R, Abshire M, Davidson PM. All Things Death and Dying: Health Professional Students Participating in the Death Cafe Model. J Palliat Med. 2018 Jun;21(6):850-852. doi: 10.1089/jpm.2017.0440. Epub 2018 Feb 2. PMID 29393728
- [Background] Rotenstein LS, Torre M, Ramos MA, Rosales RC, Guille C, Sen S, Mata DA. Prevalence of Burnout Among Physicians: A Systematic Review. JAMA. 2018 Sep 18;320(11):1131-1150. doi: 10.1001/jama.2018.12777. PMID 30326495
- [Derived] Bateman ME, Chung CH, Mascarenhas E, Hammer R, Ravindran N, Panjshiri F, Mehta P, Byrne A, Lasky S, Denson R, Brown M, Halton B, Chiurco J, Ferrell S, Ruiz B, Wentowski C, Shukla I, Bauer H, Sarma A, Bhyravabhotla K, Zu Y, Peacock E, Lefante J, Epere J, Denson JL. STOPTHEBURN: A Randomized Controlled Trial of Death Cafes for Burnout Prevention in Intensive Care Unit Employees. Ann Am Thorac Soc. 2024 Nov;21(11):1572-1582. doi: 10.1513/AnnalsATS.202312-1024OC. PMID 39052070
- [Derived] Bateman ME, Hammer R, Byrne A, Ravindran N, Chiurco J, Lasky S, Denson R, Brown M, Myers L, Zu Y, Denson JL. Death Cafes for prevention of burnout in intensive care unit employees: study protocol for a randomized controlled trial (STOPTHEBURN). Trials. 2020 Dec 11;21(1):1019. doi: 10.1186/s13063-020-04929-4. PMID 33308290